CLINICAL TRIAL: NCT07281885
Title: A Randomized Control Trial on the Efficacy of Aromatherapy in Reducing Postoperative Nausea and Vomiting in Total Joint Replacement Patients
Brief Title: Aromatherapy in Reducing PONV for Total Joint Replacement Patients
Acronym: RCT PONV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Buddhist Hospital (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Choi Wan Chan, Advanced Practice Nurse, Principal Investigator, Hong Kong Buddhist Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB-2025-242-5
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Total Joint Replacement Surgery; Postoperative Nausea and Vomiting
Keywords: Aromatherapy; PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Paralleled Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: After completion of written informed consent, participants would be randomly assigned to one of three groups (Intervention, Placebo, Control) by a designated clerical staff according to a blocked randomization list. Outcome assessors were independent, not knowing information regarding condition or grouping of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy patches (Experimental): Standard Care + Use of Aromatherapy Patches
  Interventions: Other: Aromatherapy patches
- Placebo patches (Placebo Comparator): Standard Care + Use of Placebo Patches
  Interventions: Other: Placebo Patches
- Prescribed antiemetic treatment (Active Comparator): As standard care alone
  Interventions: Drug: Control (Standard treatment)

INTERVENTIONS:
Other: Aromatherapy patches — Applying aromatherapy patch served as intervention part in addition to standard care. Aromatherapy patch will be attached to the inner side of of the patient's top covered by a plain gauze with micro-pore tape.
  Other Names: Lavender-Sandalwood patch; Orange-Ginger patch
  Arms: Aromatherapy patches
Other: Placebo Patches — On top of standard care. Placebo patch, which looks like the aromatherapy patch but contains no element of any essential oil, will be attached to the inner side of of the patient's top covered by a plain gauze with micro-pore tape.
  Arms: Placebo patches
Drug: Control (Standard treatment) — Prescribed antiemetic treatment
  Arms: Prescribed antiemetic treatment

SUMMARY:
This study investigates the effectiveness of aromatherapy in reducing postoperative nausea and vomiting (PONV) among patients undergoing total joint replacement surgery, as these complications can lead to patient discomfort and prolonged recovery. It is designed as a randomized controlled trial involving 159 participants, who will be divided into three groups: an intervention group receiving aromatherapy patches (lavender-sandalwood or orange-ginger) plus standard care, a placebo group with a placebo patch plus standard care, and a control group receiving standard care alone. PONV will be measured using the Rhodes Index of Nausea, Vomiting, and Retching (RINVR) at baseline, 30 minutes after the intervention, and every 12 hours post-surgery. Additionally, patient satisfaction will be assessed through a 5-point Likert scale survey. The primary outcome of the study is the evaluation of RINVR scores, while the secondary outcome focuses on patient satisfaction levels. Data will be statistically analyzed using two-way ANOVA for repeated measures, with a significance level defined as p < 0.05. The study aims to determine the viability of aromatherapy as a complementary treatment for PONV, potentially improving postoperative care, enhancing patient satisfaction, and offering a cost-effective alternative to conventional anti emetic treatments if proven effective.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or above
* Patients scheduled for total joint replacement surgery at the HKBH

Exclusion Criteria:

* Cognitive impairments
* Allergy to lavender, orange, ginger, or sandalwood
* Allergy to micro-pore tape
* Allergy to opioid medication
* Undergoing other therapeutic treatment for PONV control, except prescribed medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Nausea and Vomiting | Through study completion, an average of 24 hours at 4 timepoints: T0 (baseline at PACU), T1 (up to 30 minutes from applying intervention to reassessment at PACU), T2 (up to 12-hour post-intervention in ward), T3 (up to 24-hour post-intervention in ward).
  as measured by Rhodes Index of Nausea, Vomiting, and Retching, which consists of 8-item 4-point Likert-scales for nausea, vomiting, and retching symptoms with a total score ranging from 0 to 32 for each time point. The higher scores indicate the higher severity of nausea, vomiting, and retching experienced by the patient.

SECONDARY OUTCOMES:
Patient Satisfaction | Through study completion, an average of 24 hours at 4 timepoints: T0 (baseline at PACU), T1 (up to 30 minutes from applying intervention to reassessment at PACU), T2 (up to 12-hour post-intervention in ward), T3 (up to 24-hour post-intervention in ward).
  Use of patient satisfaction survey which consists of 2-item 5-point Likert scales to address the extent to which intervention could be effective in discomfort relief and control perceived by patients. The total score of the survey ranged from 2 to 10; the higher the score the more likely patients showed agreement on treatment effectiveness in discomfort relief and control.

CONTACTS AND LOCATIONS:
Overall Officials: Choi Wan CHAN, APN (NURSING), Principal Investigator — Hong Kong Buddhist Hospital
Locations (1):
- Hong Kong Buddhist Hospital, Wong Tai Sin, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bode AM, Dong Z. The Amazing and Mighty Ginger. In: Benzie IFF, Wachtel-Galor S, editors. Herbal Medicine: Biomolecular and Clinical Aspects. 2nd edition. Boca Raton (FL): CRC Press/Taylor & Francis; 2011. Chapter 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK92775/ PMID 22593941
- [Background] Chaiyakunapruk N, Kitikannakorn N, Nathisuwan S, Leeprakobboon K, Leelasettagool C. The efficacy of ginger for the prevention of postoperative nausea and vomiting: a meta-analysis. Am J Obstet Gynecol. 2006 Jan;194(1):95-9. doi: 10.1016/j.ajog.2005.06.046. PMID 16389016
- [Background] Chou FH, Avant KC, Kuo SH, Cheng HF. Assessing the psychometric and language equivalency of the Chinese versions of the Index of Nausea, Vomiting and Retching, and the Prenatal Self-Evaluation Questionnaire. Kaohsiung J Med Sci. 2005 Jul;21(7):314-21. doi: 10.1016/S1607-551X(09)70127-5. PMID 16089309
- [Background] Cardia GFE, Silva-Filho SE, Silva EL, Uchida NS, Cavalcante HAO, Cassarotti LL, Salvadego VEC, Spironello RA, Bersani-Amado CA, Cuman RKN. Effect of Lavender (Lavandula angustifolia) Essential Oil on Acute Inflammatory Response. Evid Based Complement Alternat Med. 2018 Mar 18;2018:1413940. doi: 10.1155/2018/1413940. eCollection 2018. PMID 29743918
- [Background] Ford C, Park LJ. Assessing and managing nausea and vomiting in adults. Br J Nurs. 2020 Jun 11;29(11):602-605. doi: 10.12968/bjon.2020.29.11.602. No abstract available. PMID 32516043
- [Background] Gress K, Urits I, Viswanath O, Urman RD. Clinical and economic burden of postoperative nausea and vomiting: Analysis of existing cost data. Best Pract Res Clin Anaesthesiol. 2020 Dec;34(4):681-686. doi: 10.1016/j.bpa.2020.07.003. Epub 2020 Jul 18. PMID 33288118
- [Background] A Pilot Randomized Control Trial to Assess the Impact of Lavender on Anxiety and Comfort After Cesarean Birth and the Barriers Encountered. MCN Am J Matern Child Nurs. 2022 Mar-Apr 01;47(2):E3. doi: 10.1097/NMC.0000000000000807. No abstract available. PMID 35202019
- [Background] Jin Z, Gan TJ, Bergese SD. Prevention and Treatment of Postoperative Nausea and Vomiting (PONV): A Review of Current Recommendations and Emerging Therapies. Ther Clin Risk Manag. 2020 Dec 31;16:1305-1317. doi: 10.2147/TCRM.S256234. eCollection 2020. PMID 33408475
- [Background] Marsh E, Millette D, Wolfe A. Complementary Intervention in Postoperative Care: Aromatherapy's Role in Decreasing Postoperative Nausea and Vomiting. J Holist Nurs. 2022 Dec;40(4):351-358. doi: 10.1177/08980101211065555. Epub 2021 Dec 15. PMID 34905993
- [Background] Amirshahi M, Behnamfar N, Badakhsh M, Rafiemanesh H, Keikhaie KR, Sheyback M, Sari M. Prevalence of postoperative nausea and vomiting: A systematic review and meta-analysis. Saudi J Anaesth. 2020 Jan-Mar;14(1):48-56. doi: 10.4103/sja.SJA_401_19. Epub 2020 Jan 6. PMID 31998020
- [Background] Rhodes VA, McDaniel RW. The Index of Nausea, Vomiting, and Retching: a new format of the lndex of Nausea and Vomiting. Oncol Nurs Forum. 1999 Jun;26(5):889-94. PMID 10382187
- [Background] Singh JR, Rand EB, Erosa SC, Cho RS, Sein M. Aromatherapy for Procedural Anxiety in Pain Management and Interventional Spine Procedures: A Randomized Trial. Am J Phys Med Rehabil. 2021 Oct 1;100(10):978-982. doi: 10.1097/PHM.0000000000001690. PMID 33443859
- [Background] Trambert R, Kowalski MO, Wu B, Mehta N, Friedman P. A Randomized Controlled Trial Provides Evidence to Support Aromatherapy to Minimize Anxiety in Women Undergoing Breast Biopsy. Worldviews Evid Based Nurs. 2017 Oct;14(5):394-402. doi: 10.1111/wvn.12229. Epub 2017 Apr 10. PMID 28395396